CLINICAL TRIAL: NCT03832049
Title: A Randomized, Observer-blind, Non-inferiority Trial to Evaluate Alternative Human Papillomavirus (HPV) Vaccination Schedules in Females in West Africa
Brief Title: HPV Vaccination in Africa- New Delivery Schedules Alias The HANDS HPV Vaccine Trial
Acronym: HPV
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Public Health England (Other Government); University of Cambridge (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SCC 1597
Record Dates: First submitted 2019-01-18; First posted 2019-02-06 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Human Papillomavirus Vaccine
Keywords: HPV vaccination in healthy females
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine nonavalent

STUDY DESIGN:
Intervention Model Description: a randomized, open-label, single-centre, phase 3, noninferiority clinical trial of the Gardasil 9 vaccine
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 15 to 26 years - 3 dose (Active Comparator): 9-valent human papillomavirus vaccine (Gardasil 9) - 3 doses
  Interventions: Biological: 9-valent human papillomavirus vaccine (Gardasil 9) - 3 doses
- 9 to 14 years - 2 dose (Experimental): 9-valent human papillomavirus vaccine (Gardasil 9) - 2 doses
  Interventions: Biological: 9-valent human papillomavirus vaccine (Gardasil 9) - 2 doses
- 4 to 8 years - 2 dose (Experimental): 9-valent human papillomavirus vaccine (Gardasil 9) - 2 doses
  Interventions: Biological: 9-valent human papillomavirus vaccine (Gardasil 9) - 2 doses
- 9 to 14 years - 1 dose (Experimental): 9-valent human papillomavirus vaccine (Gardasil 9) - 1 dose
  Interventions: Biological: 9-valent human papillomavirus vaccine (Gardasil 9) - 1 dose
- 4 to 8 years - 1 dose (Experimental): 9-valent human papillomavirus vaccine (Gardasil 9) - 1 dose
  Interventions: Biological: 9-valent human papillomavirus vaccine (Gardasil 9) - 1 dose

INTERVENTIONS:
Biological: 9-valent human papillomavirus vaccine (Gardasil 9) - 3 doses — 0.5mL intramuscular dose - 3 doses (0, 2 and 6 months)
  Arms: 15 to 26 years - 3 dose
Biological: 9-valent human papillomavirus vaccine (Gardasil 9) - 2 doses — 0.5mL intramuscular dose - 2 doses (0 and 6 months)
  Arms: 4 to 8 years - 2 dose; 9 to 14 years - 2 dose
Biological: 9-valent human papillomavirus vaccine (Gardasil 9) - 1 dose — 0.5mL intramuscular dose - 1 doses (0 months)
  Arms: 4 to 8 years - 1 dose; 9 to 14 years - 1 dose

SUMMARY:
A randomized, observer-blind non-inferiority trial to evaluate alternative human papillomavirus (HPV) vaccination schedules in young females in West Africa.

DETAILED DESCRIPTION:
This study is a randomized, open-label, single-centre, phase 3 non-inferiority clinical trial of the Gardasil 9 vaccine. It will be undertaken in three female cohorts (15 to 26 years old; 9 to 14 years-olds and 4 to 8 year-olds). In total 1720 female participants will be recruited in a rural setting in The Gambia, West Africa.

The Gardasil 9 vaccine is a recombinant L 1 VLP vaccine containing HPV types 6, 11,16,18,31,33,45,52 and 58 VLP. It is licensed by both European Medicines Agency and the US Food and Drug Administration as a two or three dose schedule to 9 to 14 year olds and as a three dose schedule to 15 to 26 years olds. The license covers both males and females. The vaccine is not currently licensed for those under 9 years of age and it is not licenced in The Gambia.

All females within the 15 to 26 year-old cohort will receive three doses of Gardasil 9 at 0, 2 and 6 months and represent the reference group for the purposes of the serological non-inferiority analysis. This is the only group for which efficacy data for the vaccine are available. Females in the 9 to 14 year old and 4 to 8 year old cohorts will be randomized to receive either one or two doses of Gardasil 9. In both groups, the two doses will be administered at 0 and 6 months.

The primary and secondary immunogenicity objectives will be analysed based on serological Samples taken 4 to 6 weeks after the last dose of vaccine received according to group. Additional analysis will be undertaken at 12, 24 and 36 months. The Sampling schedule is aligned with the schedule in other immunogenicity trials to facilitate comparison and potential immunobridging to future one-dose efficacy data. In addition, the stability of the antibody concentrations between 12 and 24 and again between 24 and 36 months according to schedule and age-group aims to allow longer term predictions regarding the maintenance of antibody concentration to be made.

A Sub-study will be undertaken within the main trial to compare in detail early immunological events taking place following Gardasil 9. The quantitative and qualitative changes in these events following a first and following subsequent doses of the vaccine and also according to age will be assessed and related to the early and long-term antibody concentrations induced by the vaccine. There are currently no data exploring the basis for the progressive increase in the immunogenicity of the HPV vaccines apparent with decreasing age. These may have their origins in the early innate response following vaccination-which will be assessed at a cellular as well as transcriptomic level, as well as in the subsequent adaptive profile.

Similarly, the cellular basis for the sustained seropositivity induced by the HPV vaccines even apparent following a single vaccine dose is little understood. The window onto which plasmablasts and memory B-cell populations in the circulation is transient following vaccination. However, enumerating and characterizing these populations and relating them in the same way to early and long term antibody concentration aims to provide insight into the relative roles of these populations and how they are influenced by the age of the vaccine and the number of vaccine doses received.

Individuals in the sub-study will contribute serological data to the main trial and will be followed up in the same way but will be consented for one additional blood sample after each vaccination. Up to 120 participant in each group in the main trial will be randomized to groups A, B or C, with 40 participants in each of these groups. This number aims to generate a dataset of at least 30 analyzable individuals per schedule and age group.

ELIGIBILITY:
Inclusion Criteria:

* Signed/thumb-printed informed consent obtained from the participant's parent (4 to 17 year-olds) or signed/thumb-printed informed consent obtained from the participant (18 years and above)
* Signed/thumb-printed assent obtained from the participant (12 to 17 year-olds only).
* Documented verbal assent obtained from the participant (6 to 11 year-olds only)
* Participant is of female sex (based on participant/parent self-report)
* Participant is between 4 and 26 years of age inclusive
* Parent/participant is willing and judged able to comply with the necessary study procedures
* Parent/participant does not have established plans to leave the study area for a prolonged period/indefinitely during the 3 year follow-up period
* Participant is resident within the study area (no fixed boundaries will be set and decisions will be made on a case-by-case basis by the study team taking into account not only distance but also transport links, accessibility for the purposes of safety data collection, willingness of the parent/participant to travel)
* Place of residence of the participant must be readily identifiable

Exclusion Criteria:

* Receipt of other investigational medicinal products (IMP) in a period of 12 months prior to the day of randomization and vaccination or plans to receive IMP during the trial.
* Presence of significant chronic health problems requiring long-term medication or medical follow-up including respiratory, cardiac, gastrointestinal, hepatic, renal, neurological, musculoskeletal, haematological or other conditions based on parental history and physical examination of the participant. Participants with known sickle cell disease (but not sickle cell trait) will be excluded.
* History of severe allergic reactions to any prior vaccine or to any component of the study vaccine (including alum (amorphous aluminum hydroxyphosphate sulphate), yeast or Benzonase). Severe allergic reactions are defined as reactions requiring urgent medical intervention including reactions with any degree of cardiorespiratory compromise. The occurrence of a mild rash without other associated symptoms or signs does not generally represent an exclusion. Allergic reactions should be distinguished from the local and systemic reactogenicity expected in the first few days following vaccination which is not an exclusion to vaccination
* Prior receipt of an HPV vaccine
* Receipt of any vaccine in the 28 days prior to randomization and vaccination‡
* History of thrombocytopenia or coagulation disorders which represent contraindications in intramuscular (IM) vaccination
* Known congenital or acquired immune deficiency or history strongly indicative of abnormal immune function. HIV testing will not be undertaken as part of the routine screening procedures due to the relatively low prevalence of HIV expected in the population (~1-3%) and the established safety and immunogenicity profile of Gardasil in HIV positive individuals.
* Receipt of medications or other treatments known to suppress the immune system in a period of 12 months prior to the day of randomization or plans to receive such medications and treatments during the course of the trial. Such medications and treatments include but not limited to high dose non-replacement) oral or parenteral steroids for more than 14 days, chemotherapeutic agents, methotrexate, cyclophosphamide, cyclosporin, Tacrolimus, any monoclonal antibody therapy and radiotherapy. The use of topical and inhaled steroids are not exclusion criteria.
* Receipt of intravenous immunoglobulins or blood products within a period of 12 months prior to the day of randomization and vaccination or plans to receive such products during the course of the trial.
* Pregnancy (females in the 15 to 26 years old cohort will require a urine pregnancy test as part of the screening procedures and will also have a urine pregnancy test undertaken prior to the second and third vaccination and vaccination delayed if pregnancy is confirmed. A minimum of 42 days from the end of pregnancy (irrespective of outcome) will be left before the delayed vaccination is administered. Participants who are pregnant at initial screening will not be re-screened but will be defined as screen failures. Breast feeding is not an exclusion criterion
* Intention to become pregnant within six months of enrollment in the trial. Confirmation regarding the use of a reliable method of contraception is not required but females who are actively seeking to become pregnant within six months of enrollment will be excluded.
* Fever (>38.0°C) on the day of vaccination or documented fever (>38.0°C) within the 24 hours preceding vaccination
* Abnormal (Grade > 1) vital signs (heart rate, respiratory rate, blood pressure) on the day of vaccination
* Positive rapid diagnostic test (RDT) or blood film for malaria on the day of vaccination
* Clinically-significant (Grade > 2) acute illness present on the day of vaccination (minor illnesses including upper respiratory tract infections, diarrhoeal illness and skin complaints not associated with fever or significant systemic upset are not in themselves reasons for exclusion)

Ages: 4 Years to 26 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Participant is of female sex (based on participant/parent self-report)
Enrollment: 1720 (Actual)
Dates: Start 2019-09-14 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Antibodies measured by 9-valent HPV competitive Luminex immunoassay (cLIA) (mMU/mL) | 4 weeks after last vaccine dose
  HPV types, 6, 11, 16, 18, 31, 33, 45, 52 and 58
Acute allergic reaction (Grade 0 - 4) | Day of vaccination (day 0)
  Solicited systemic reactogenicity recorded in 4 to 8 year olds and 9 to 14 year olds
Injection site pain (Grade 0 - 4) | Days 0 to 6 after vaccination
  Solicited local reactogenicity recorded in 4 to 8 year olds and 9 to 14 year olds
Injection site redness (Grade 0 - 4) | Days 0 to 6 after vaccination
  Solicited local reactogenicity recorded in 4 to 8 year olds and 9 to 14 year olds
Injection site swelling (Grade 0 - 4) | Days 0 to 6 after vaccination
  Solicited local reactogenicity recorded in 4 to 8 year olds and 9 to 14 year olds
Injection site pruritus (Grade 0 - 4) | Days 0 to 6 after vaccination
  Solicited local reactogenicity recorded in 4 to 8 year olds and 9 to 14 year olds
Temperature in degrees Centigrade | Days 0 to 6 after vaccination
  Recorded in 4 to 8 year olds and 9 to 14 year olds
Nausea/vomiting (Grade 0 - 4) | Days 0 to 6 after vaccination
  Solicited systemic reactogenicity recorded in 4 to 8 year olds and 9 to 14 year olds
Headaches (Grade 0 - 4) | Days 0 to 6 after vaccination
  Solicited systemic reactogenicity recorded in 4 to 8 year olds and 9 to 14 year olds
Dizziness (Grade 0 - 4) | Days 0 to 6 after vaccination
  Solicited systemic reactogenicity recorded in 4 to 8 year olds and 9 to 14 year olds
Fatigue (Grade 0 - 4) | Days 0 to 6 after vaccination
  Solicited systemic reactogenicity recorded in 4 to 8 year olds and 9 to 14 year olds
Myalgia/arthralgia (Grade 0 - 4) | Days 0 to 6 after vaccination
  Solicited systemic reactogenicity recorded in 4 to 8 year olds and 9 to 14 year olds
Unsolicited adverse event (AE) including serious adverse events | Day 0 to day 28 following each vaccination
  Unsolicited AE will be recorded in 4 to 8 years olds and 9 to 14 year olds
Suspected unexpected serious adverse reactions (SUSAR) | Day 0 to month 36
  SUSAR will be collected from all participants

SECONDARY OUTCOMES:
Antibodies measured by 9-valent HPV cLIA (mMU/mL) | 12 months after first vaccination
  HPV types, 6, 11, 16, 18, 31, 33, 45, 52 and 58
Antibodies measured by 9-valent HPV cLIA (mMU/mL) | 24 months after first vaccination
  HPV types, 6, 11, 16, 18, 31, 33, 45, 52 and 58
Antibodies measured by 9-valent HPV cLIA (mMU/mL) | 36 months after first vaccination
  HPV types, 6, 11, 16, 18, 31, 33, 45, 52 and 58
Antibodies measure by 9-valent HPV total IgG (TIgG) | 4 weeks after last vaccine dose
  HPV types, 6, 11, 16, 18, 31, 33, 45, 52 and 58
Antibodies measure by 9-valent HPV TIgG | 12 months after first vaccination
  HPV types, 6, 11, 16, 18, 31, 33, 45, 52 and 58
Antibodies measure by 9-valent HPV TIgG | 24 months after first vaccination
  HPV types, 6, 11, 16, 18, 31, 33, 45, 52 and 58
Antibodies measure by 9-valent HPV TIgG | 36 months after first vaccination
  HPV types, 6, 11, 16, 18, 31, 33, 45, 52 and 58

CONTACTS AND LOCATIONS:
Overall Officials: Ed Clarke, MB ChB PhD, Principal Investigator — Medical Research Council @ LSHTM
Locations (1):
- Ed Clarke, Banjul, Outside U.S. and Canada, The Gambia

REFERENCES:
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263